CLINICAL TRIAL: NCT00006239
Title: A Phase I, Dose-Finding Trial of Sodium Phenylbutrate (NSC 657802) in Combination With All Trans-retinoic Acid (ATRA, NSC 122758) in Patients With Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML)
Brief Title: Phenylbutyrate and Tretinoin in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: J9879 CDR0000068164; R01CA067803 (NIH); P30CA006973 (NIH); JHOC-J9879; JHOC-99072306; NCI-T98-0068
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; previously treated myelodysplastic syndromes; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Congenital Abnormalities | interventions — 4-phenylbutyric acid; Tretinoin

INTERVENTIONS:
Drug: sodium phenylbutyrate
Drug: tretinoin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Tretinoin may help hematologic cancer cells develop into normal white blood cells.

PURPOSE: Phase I trial to study the effectiveness of combining phenylbutyrate and tretinoin in treating patients who have hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and toxicity of phenylbutyrate and tretinoin in patients with myelodysplastic syndromes, chronic myelomonocytic leukemia, or acute myeloid leukemia.
* Determine the pharmacokinetic interaction of this regimen in these patients.
* Determine any potential therapeutic activity of this regimen in these patients.

OUTLINE: This is a dose escalation study of tretinoin.

Patients receive phenylbutyrate IV continuously on days 1-7 of weeks 1, 5, 7, 9, 11, 13, 15, 17, and 19. Patients also receive oral tretinoin three times daily on days 1-7 of weeks 3, 5, 7, 9, 11, 13, 15, 17, and 19. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of tretinoin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 6 patients experience dose limiting toxicities.

An additional cohort of 6 patients is accrued at the MTD. These patients receive phenylbutyrate IV continuously on days 1-3 of weeks 1 and 3-18. These patients also receive oral tretinoin three times daily on days 1-3 of weeks 2-18. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed myelodysplastic syndrome (MDS)

  * Refractory anemia
  * Primary refractory leukopenia or thrombocytopenia with morphologic features of MDS
  * Refractory anemia with excess blasts (RAEB)
  * Refractory anemia with ringed sideroblasts
  * RAEB in transformation
  * Must have excess blasts or be hematopoietically compromised, defined as one of the following:

    * RBC transfusion dependent
    * Granulocyte count less than 1,000/mm^3
    * Platelet count less than 50,000/mm^3 OR
* Diagnosis of chronic myelomonocytic leukemia

  * Hematopoietically compromised (as defined above) OR
  * Excess blasts OR
  * Evaluable disease related symptomatology (organomegaly or leukemia cutis) OR
* Diagnosis of acute myeloid leukemia

  * WBC less than 20,000/mm^3 and stable for at least 2 weeks
  * Unlikely to require cytotoxic therapy during study
* No CNS or pulmonary leukostasis or CNS leukemia

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics
* Hemoglobin at least 8 g/dL (transfusion allowed)
* No disseminated intravascular coagulation

Hepatic:

* Bilirubin less than 2.0 mg/dL (unless due to hemolysis or Gilbert's syndrome)

Renal:

* Creatinine less than 2.0 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 2 weeks prior, during, and for 3 months after study
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 3 weeks since prior biologic therapy, including hematopoietic growth factors, and recovered

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks (1 month for MDS patients) since prior chemotherapy and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 3 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Primary Completion 2005-02 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven D. Gore, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States